CLINICAL TRIAL: NCT07304206
Title: Comparison of the Effects of Three Different Anesthetic Methods on Postoperative Agitation in Septoplasty Surgery
Brief Title: The Effects of Three Different Anesthetic Methods on Postoperative Agitation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ülkü Özgül, Prof.Dr., Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CIVIA Septoplasty
Record Dates: First submitted 2025-12-01; First posted 2025-12-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Emergence Agitation; Septoplasty Surgeries
Keywords: anesthesia; emergence agitation; tiva
MeSH Terms: conditions — Emergence Delirium | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participant: The participant will be unaware of which anesthesia method is performed in the perioperative period.
  Care Provider: The second anesthesiologist will wake the patient after the anesthesia has been terminated and will not know which anesthesia method was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group S (Sevoflurane) (Active Comparator): After entering the patient's demographic data (height, gender, weight, and age), the initial target concentration (Ce) at the site of action for propofol will be recorded as 4 µg/mL in the Eleveld model (MedCaptain Eleveld HP TCI Infusion Syringe Pump), and the target concentration (Ce) for remifentanil will be recorded as 4 ng/mL in the Minto model. Ventilation will be performed with a face mask using 100% O2 after loss of consciousness and disappearance of the eyelash reflex. When the BIS value drops below 60, measurement of the degree of neuromuscular blockade (TOFWatch S monitor; Organon, Dublin, Ireland) will be initiated. Rocuronium will be administered as a bolus at a dose of 0.6 mg/kg according to ideal body weight, followed by intubation. Anesthesia maintenance will be provided with sevoflurane to keep the BIS value between 40-60. The target remifentanil concentration will be increased or decreased by 0.5 ng/mL to maintain mean arterial pressure (MAP) at 60-70 mmHg.
  Interventions: Drug: SEVOFLURANE
- Group T (TIVA) (Active Comparator): After entering the patient's demographic data (height, gender, weight, and age), the Eleveld model (MedCaptain Eleveld HP TCI Infusion Syringe Pump) will be set to Ce 4 µg/mL for propofol and Ce 4 ng/mL for remifentanil in the Minto model. Ventilation with a face mask will be performed using 100% O2 after loss of consciousness and disappearance of the eyelash reflex. When the BIS value drops below 60, measurement of the degree of neuromuscular blockade (TOF - watch TOFWatch SX, Organon, Ireland) will be initiated. Rocuronium will be administered as a bolus at a dose of 0.6 mg/kg according to ideal body weight, and intubation will be performed. Anesthesia will be maintained by increasing or decreasing the target concentration of propofol by 0.5 μg/mL to keep the BIS value in the 40-60 range. The target remifentanil concentration will be increased or decreased by 0.5 ng/mL to maintain mean arterial pressure at 60-70 mmHg.
  Interventions: Drug: TIVA
- Group C (CIVIA) (Active Comparator): After entering the patient's demographic data (height, gender, weight, and age), the Ce level will be set to 4 µg/mL for propofol in the Eleveld model and 4 ng/mL for remifentanil in the Minto model. Ventilation will be performed with a face mask using 100% O2 after loss of consciousness and disappearance of the eyelash reflex. When the BIS value drops below 60, measurement of the degree of neuromuscular blockade will be initiated. Rocuronium will be administered as a bolus at a dose of 0.6 mg/kg according to ideal body weight, and intubation will be performed. For maintenance of anesthesia, inhaled sevoflurane concentration will be started at 0.5 MAC, while the propofol Ce level will be adjusted to 2 µg/mL, and propofol will be increased or decreased by 0.5 μg/mL to maintain the BIS target in the 40-60 range. Remifentanil infusion will be administered to maintain mean arterial pressure at 60-70 mmHg, with a titration of 0.5 ng/mL.
  Interventions: Drug: CIVIA

INTERVENTIONS:
Drug: SEVOFLURANE — Anesthetic management will be made with sevoflurane
  Arms: Group S (Sevoflurane)
Drug: TIVA — Propofol and remifentanil will be given with TCİ device for anesthetic induction and management
  Arms: Group T (TIVA)
Drug: CIVIA — In this group patients <0.5 MAC sevoflurane will be used in combination with total intraveous method (This method described above )
  Arms: Group C (CIVIA)

SUMMARY:
Adult patients undergoing septoplasty surgery will be evaluated in this study. The three different anesthesia methods used will be examined for psotoperative agitation: Total intravenous anesthesia (TIVA), Combined anesthesia with sevoflurane and intravenous agents (sevoflurane-CIVIA), Balanced inhalation anesthesia with sevoflurane. Recovery patterns is extubation time, eye opening time, emergence agitation, postoperative nausea and vomiting and postoperative recovery unit discharge time.

DETAILED DESCRIPTION:
Agitation, defined as restlessness, disorientation, arousal, and/or inconsolable crying, is a common phenomenon seen in the early phase of recovery from general anesthesia. It can lead to respiratory depression, nausea, and vomiting, as well as increases in blood pressure, heart rate, and myocardial oxygen consumption. Hypoxia can lead to serious complications such as aspiration pneumonia, bleeding, or reoperation. Although its pathogenesis remains unclear, ear, nose, and throat (ENT) surgical procedures have been reported to have a higher incidence of agitation in both adults and children.

Classic general anesthesia is performed with induction using an intravenous hypnotic such as propofol and maintenance with a volatile anesthetic such as sevoflurane, along with intermittent or continuous opioids and muscle relaxants. Opinions differ regarding the effects of inhalational and intravenous anesthesia on maintenance. A 2015 retrospective study investigating the risk factors for emergence agitation after rhinoplasty reported that sevoflurane use more than doubled the risk of emergence agitation.

The use of propofol and sevoflurane for maintenance has recently been recommended due to the antiemetic effects of propofol, the myocardial protective effects of sevoflurane, and the potential for smoother emergence from the administration of small amounts of each anesthetic . This study aimed to compare the occurrence of emergence agitation after inhalation anesthesia, total intravenous anesthesia with TCI, and combined inhalation and intravenous anesthesia in patients undergoing septoplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years old.
* American Society of Anesthesiologists (ASA) Physical Status Class I or II.
* Scheduled for elective septoplasty surgery.
* Scheduled to receive general anesthesia

Exclusion Criteria:

* History of revision septoplasty
* Known allergy to nonsteroidal anti-inflammatory drugs (NSAIDs) or the study drugs
* History of bleeding disorder
* History of allergy
* ASA Physical Status greater than III
* Body Mass Index (BMI) $> 30
* History of hypertension, cardiovascular diseases, or cerebrovascular diseases
* History of renal dysfunction
* Use of psychiatric medications
* History of substance abuse
* Patients who refuse to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Emergence agitation | Immediately after tracheal extubation
  Emergence agitation will be assessed using the Richmond Agitation-Sedation Scale (RASS). RASS is a 10-point scale ranging from +4 to -5, measures agitation, sedation level, and responsiveness.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting (PONV) | Immediately post-op, 15 minutes, and 30 minutes in the Post-Anesthesia Care Unit (PACU)
  Postoperative nausea and vomiting assessed on a 4-point scale:
  None: 0 Mild nausea: 1 Moderate nausea: 2 Frequent vomiting: 3 Severe vomiting: 4
Extubation time | Immediately postoperative period
  The time when patients are extubated after all anesthetic drugs have been discontinued
Recovery time | Continuous observation for 30 minutes in the PACU.
  Recovery time is between the termination of anesthesia and the patient being discharged from the postoperative recovery room (PACU) with an Aldrete score of >9.

CONTACTS AND LOCATIONS:
Overall Officials: Ülkü Özgül, Professor, Study Director — turgut özal medical center Department of Anesthesiology and Reanimation
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wolf A, Selpien H, Haberl H, Unterberg M. Does a combined intravenous-volatile anesthesia offer advantages compared to an intravenous or volatile anesthesia alone: a systematic review and meta-analysis. BMC Anesthesiol. 2021 Feb 15;21(1):52. doi: 10.1186/s12871-021-01273-1. PMID 33588751